CLINICAL TRIAL: NCT04922905
Title: Nervous System Symptoms Associated With COVID 19 : NS-COV
Brief Title: Nervous System Symptoms Associated With COVID 19
Acronym: NS-COV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RC31/20/0178
Record Dates: First submitted 2021-06-09; First posted 2021-06-11 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: Nervous system; coronavirus; SARS-CoV-2; Nervous system symptoms
MeSH Terms: conditions — COVID-19; Neurologic Manifestations; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: This is an observational, prospective, cross-sectional and monocentric cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEURO + (Other): Patients "neuro +" are those with a CASE score ≥ 2, "Neuro +" patients will benefit from additional evaluations using paraclinical examinations
  Interventions: Other: NEURO +
- NEURO - (Other): Patients "neuro -" are those with a CASE score < 2
  Interventions: Other: NEURO -

INTERVENTIONS:
Other: NEURO + — The participants will undergo several questionnaires after their classic clinical evaluation allowing to determine the Clinical Assessment Scale in Autoimmune Encephalitis (CASE) score :
  * The dissociative peri-traumatic experiences questionnaire (Birmes et al., 2005)
  * the Peri traumatic distress inventory (Jehel et al., 2005)
  * and the Shortness, Trembling, Racing, Sweating (STRS) (Bracha et al., 2004)
  Neuro + patients will also have a Brain MRI, cerebrospinal fluid analysis, EEG, as well as an ambulatory sleep recording and electromyography depending on the symptoms observed.
  Arms: NEURO +
Other: NEURO - — The participants will undergo several questionnaires after their classic clinical evaluation allowing to determine the Clinical Assessment Scale in Autoimmune Encephalitis (CASE) score :
  * The dissociative peri-traumatic experiences questionnaire (Birmes et al., 2005)
  * the Peri traumatic distress inventory (Jehel et al., 2005)
  * and the Shortness, Trembling, Racing, Sweating (STRS) (Bracha et al., 2004)
  Arms: NEURO -

SUMMARY:
This study aim to prospectively evaluate the neuropsychiatric symptoms of patients infected with the SARS-CoV-2 virus by a standardized neuropsychiatric examination : the global CASE scale (Clinical Assessment Scale in Autoimmune Encephalitis), and the prevalence of disturbances of consciousness, focal neurological deficit, cognitive impairment, headache, anosmia, sleep disturbances, impaired autonomic nervous system and peritraumatic stress.

ELIGIBILITY:
Inclusion Criteria:

* Being hospitalized at the Toulouse University Hospital for a COVID-19 infection proven by a probable PCR or COVID-type examination on the chest scan
* Have given oral consent for the collection of clinical neurological data
* Be in a clinical state compatible with a 30-minute neurological examination
* Be French-speaking
* Be affiliated to a Social Security scheme

Exclusion Criteria:

* Refusal of the neurological examination
* History of neurological pathology at a severe stage
* Pregnant or breastfeeding woman
* Persons with tutors or curators

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
percentage of patients in the Neuro + and Neuro- groups | Baseline T0 : inclusion visit
  The percentage is deducted from the score on a global scale by the Clinical Assessment Scale in Autoimmune Between 0 and 1, patients will be classified in the Neuro group, if this score is greater than or equal to 2, patients will be classified in the Neuro + group.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Rafiq, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No